CLINICAL TRIAL: NCT02680639
Title: The Use of High Frequency Oscillations With Noninvasive Ventilation (NIV) in Hypercapnic Chronic Obstructive Pulmonary Disease (COPD) Participants
Brief Title: The Use of High Frequency Oscillations With NIV in Hypercapnic COPD Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had a high screen fail rate, enrollment was open over a year, only 3 completed.
Sponsor: Philips Respironics (Industry)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: HRC-1433-HFO-SS
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: High-Frequency Ventilation; Biphasic Continuous Positive Airway Pressure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- optimal EPAP determination (Active Comparator): On the BiPAP Synchrony ventilator the EPAP (and IPAP) will be automatically adjusted by the ventilator to find optimal EPAP that abolishes EFL. Peak-to-Peak pressure oscillations will be set at 2.5 cmH2O (centimeters of water)
  Interventions: Device: BiPAP Synchrony ventilator
- Optimized EPAP w/ no peak-to-peak (Experimental): On the BiPAP Synchrony ventilator the EPAP (and IPAP) will be set at optimal pressure as determined by the Auto EPAP. Peak-to-Peak pressure oscillations will be set at 0 cmH2O (centimeters of water)
  Interventions: Device: BiPAP Synchrony ventilator
- Optimized EPAP w/ max peak-to-peak (Experimental): On the BiPAP Synchrony ventilator EPAP (and IPAP) will be set at optimal pressure as determined by the Auto EPAP. Peak-to-Peak pressure oscillations will be set at 5 cmH2O (centimeters of water)
  Interventions: Device: BiPAP Synchrony ventilator
- non-optimized EPAP w/ no peak-to-peak (Experimental): On the BiPAP Synchrony ventilator EPAP will be set at 4 cmH2O and IPAP will be set at 10 cmH2O (centimeters of water). Peak-to-Peak pressure oscillations will be set at 0 cmH2O (centimeters of water).
  Interventions: Device: BiPAP Synchrony ventilator

INTERVENTIONS:
Device: BiPAP Synchrony ventilator — The BiPAP Synchrony ventilator will be used to determine Expiratory Positive Airway Pressure (EPAP). The ventilator will be used with varying pressure supports and oscillations depending on what arm of the study the participant is in.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of chronic morbidity and mortality throughout the world, being the fourth leading cause of death in the world.

This study is designed to detect COPD participants with Expiratory Flow Limitation. EFL occurs when the airways become compressed which usually results when a pressure outside the airway exceeds the pressure inside the airway.

Participants will undergo study eligibility procedures at visit 1. At visit 2 participants will undergo a baseline auto-EPAP (Expiratory Positive Airway Pressure) measurement. Then the order will be randomized to three different treatment methods. Between each treatment there will be at least a 10 minute washout period in order for CO2 to stabilize and return to baseline.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of chronic morbidity and mortality throughout the world, being the fourth leading cause of death in the world.

COPD is a disease that results in varying degrees of dyspnea, or shortness of breath. Spirometry is a method of diagnosing COPD with the presence of a post bronchodilator FEV1 <80% of the predicted value in combination with an FEV1 / FVC <70%. This would confirm that there is a presence of airflow limitation that is not fully reversible.

The presence of airflow limitation has been identified as one of the main causes of dyspnea in patients with chronic obstructive pulmonary disease (1). Expiratory Flow Limitation (EFL) occurs when the airways become compressed which usually results when a pressure outside the airway exceeds the pressure inside the airway. As an airflow obstruction worsens, EFL appears at much lower flows for a given lung volume and it becomes present at rest or at least develops early during exercise (2).

Early detection of EFL consisted of either invasive balloon catheterization or relatively complex plethysmographic techniques. An alternative approach, and one that will be used in this study, involves utilizing the Forced Oscillation Technique (FOT).

Alternatively High Frequency Oscillations (HFO) has shown to effectively lower CO2 levels, but traditionally require intubation or a trans tracheal catheter. Treatment with a specialized noninvasive ventilator is possible and it is proposed that therapy can be augmented by the application of an optimized EPAP to splint open the lower airways in order to increase the diffusive capabilities of the high frequency oscillations into lower alveolar regions. There are approximately 25 million hypercapnic patients with EFL that could benefit from this therapy. High frequency oscillations integrated into a specialized noninvasive ventilator has the advantages of lower cost than other solutions and significantly lower medical risks. In addition, high frequency oscillation uses lower pressures to achieve effective therapy which means less chance of barotrauma and greater patient acceptance.

This study will enroll subjects at a screening visit. Screening will include a physical exam and vital signs, pregnancy test (if applicable), questionnaires, pulse oximetry, measure of carbon dioxide levels, determination of EFL by an auto- Expiratory Positive Airway Pressure (EPAP) ventilator, and spirometry.

If the patient is eligible and tolerates the above procedures, they will be asked to complete an in home-based sleep study prior to visit 2. Alice Night One/ Alice PDX are portable home sleep testing devices that record information about breathing.

At visit 2 participants will be monitored continuously via a 3 lead EKG, oxygen saturation by pulse oximetry (SPO2), Carbon Dioxide concentration(TcCO2) monitor, RespiTrace belt and ventilator data.

During Visit 2, participants will first undergo a repeat optimal EPAP determination and then trial 3 different sessions of High Frequency Oscillation (HFO) therapy for 20 minutes with at least a 10 minute wash out period between each session to allow the participant's CO2 to stabilize or return to baseline. The order of the sessions will be randomized for each patient. Participants will be placed in a semi-recumbent position and wear a nasal CPAP mask for each session. A TcCO2 monitor patch will be placed on the skin (forehead area) to collect carbon dioxide measurements during each session. A RespiTrace belt will placed on the participants' chest wall to measure chest wall and diaphragmatic excursion during each session. A 3 lead EKG will also be used to monitor cardiac activity during each session.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years of age; < 85 years of age
* Participants that have been physician diagnosed (primary diagnosis) with Obstructive Airway Disease (to include:Chronic Obstructive Pulmonary Disease (COPD); Bronchiectasis; Severe Asthma); forced expiratory volume in 1 second (FEV1) < 60% FEV1/ forced vital capacity (FVC) <60%
* Arterial CO2 > 45 mmHg as determined by blood gas (PaCO2) or transcutaneous (tcCO2) >50 within the past month
* Ability to provide consent
* Participant has not used Non-Invasive Ventilation (BiPAP/CPAP) therapy in the past 8 hours
* Participant has no child bearing potential OR a negative pregnancy test in a woman of childbearing potential

Exclusion Criteria:

* Participants that have not returned to their baseline health status from an exacerbation of COPD or other pulmonary problems or have not established at least two weeks of stability at a new baseline.
* Use of antibiotics or prednisone for a COPD exacerbation within the previous 4 weeks.
* Uncontrolled Hypertension
* Participants that require greater than 3 liters of oxygen at rest
* History of cardiovascular instability, including uncontrolled ventricular arrhythmias, angina, diastolic BP > 100 mmHg and all Participants with pacemakers
* Any major non-COPD uncontrolled disease or condition, such as congestive heart failure, malignancy, end-stage heart disease, liver or renal insufficiency (that requires current evaluation for liver or renal transplantation or dialysis), amyotrophic lateral sclerosis, or severe stroke, or other condition as deemed appropriate by investigator as determined by review of medical history and / or participant reported medical history
* History of pneumothorax
* Apnea Hypopnea Index (AHI) > 15 via in-home sleep study
* Excessive alcohol intake (> 6oz hard liquor, 48 oz. beer or 20 oz. wine daily), or illicit drug use by review of medical history and / or participant reported medical history
* Daily use of prescribed narcotics (greater than 30 mg morphine equivalent)
* History of Giant bullous emphysema
* A positive urine pregnancy test when screening for study

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sciurba, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD), only aggregate data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were in enrolled from a single site in Pittsburgh PA. The study opened Mid 2015 with first enrollment November 2015 and continued into August 2016.
Groups:
- Screening Period: All study participants that were consented to the study.
- Optimal, Optimized P2P, Non-Optimized NP2P, Optimized NP2P; Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized NP2P: Optimal - optimal EPAP determination first, Optimized P2P - Optimized EPAP w/ max peak-to-peak second, Non-Optimized NP2P - non-optimized EPAP w/ no peak-to-peak third, and Optimized NP2P - Optimized EPAP w/ no peak-to-peak last
Period: Screening Period
Arm/Group | Screening Period | Optimal, Optimized P2P, Non-Optimized NP2P, Optimized NP2P | Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized NP2P
Started | 10 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Screen Failure | 7 | 0 | 0
Period: High Frequency Oscillation (HFO) Therapy
Arm/Group | Screening Period | Optimal, Optimized P2P, Non-Optimized NP2P, Optimized NP2P | Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized NP2P
Started | 0 | 2 | 1
Completed | 0 | 2 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that signed consent.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Carbon Dioxide Levels
Description: Transcutaneous carbon dioxide (TcCO2) monitoring is a non-invasive alternative to arterial blood sampling. Carbon Dioxide Levels will be measured for each participant as they complete each arm.
Time Frame: Baseline and 20 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Optimal EPAP Determination: On the BiPAP Synchrony ventilator the EPAP (and IPAP) will be automatically adjusted by the ventilator to find optimal EPAP that abolishes expiratory flow limitation (EFL). Peak-to-Peak pressure oscillations will be set at 2.5 cmH2O (centimeters of water)
  BiPAP Synchrony ventilator: The BiPAP Synchrony ventilator will be used to determine Expiratory Positive Airway Pressure (EPAP). The ventilator will be used with varying pressure supports and oscillations depending on what arm of the study the participant is in.
- Non-optimized EPAP w/ no Peak-to-peak: On the BiPAP Synchrony ventilator EPAP will be set at 4cmH2O and IPAP will be set at 10cmH2O (centimeters of water). Peak-to-Peak pressure oscillations will be set at 0 cmH2O (centimeters of water).
  BiPAP Synchrony ventilator: The BiPAP Synchrony ventilator will be used to determine Expiratory Positive Airway Pressure (EPAP). The ventilator will be used with varying pressure supports and oscillations depending on what arm of the study the participant is in.
Arm/Group | Optimal EPAP Determination | Optimized EPAP w/ no Peak-to-peak | Optimized EPAP w/ Max Peak-to-peak | Non-optimized EPAP w/ no Peak-to-peak
Number analyzed (Participants) | 3 | 3 | 3 | 3
mmHg
  Baseline | 57.8 (9.1) | 52.6 (7.1) | 53.1 (9.8) | 52.4 (8.5)
  20 Minutes | 51.1 (8.7) | 49.7 (6.0) | 50.2 (8.5) | 49.7 (8.3)

2. Secondary Outcome: Respiratory Rate
Description: Minute ventilation in regards to respiratory rate and volume of gas exchanged will be measured for each participant as they complete each arm.
Time Frame: 20 minutes
Population: Respiratory rate was not able to be obtained for one participant.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Optimal EPAP Determination | Optimized EPAP w/ no Peak-to-peak | Optimized EPAP w/ Max Peak-to-peak | Non-optimized EPAP w/ no Peak-to-peak
Number analyzed (Participants) | 2 | 2 | 2 | 2
breaths per minute | 18.5 (2.5) | 22 (3) | 23 (2) | 24 (0)

3. Secondary Outcome: Tidal Volume
Description: Minute ventilation in regards to volume of gas exchanged will be measured for each participant as they complete each arm.
Time Frame: 20 minutes
Population: Tidal volume was not able to be obtained for one participant.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Optimal EPAP Determination | Optimized EPAP w/ no Peak-to-peak | Optimized EPAP w/ Max Peak-to-peak | Non-optimized EPAP w/ no Peak-to-peak
Number analyzed (Participants) | 2 | 2 | 2 | 2
mL | 373 (77) | 272.5 (29.5) | 293 (26) | 253 (24)

4. Secondary Outcome: Minute Ventilation for Carbon Dioxide
Description: Minute Ventilation in regards to the diffusion state of the lungs and carbon dioxide will be measured for each participant as they complete each arm.
Time Frame: 20 minutes
Population: Respiratory rate and Tidal volume were not able to be obtained for one participant. Therefore minute ventilation was not able to be calculated.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Optimal EPAP Determination | Optimized EPAP w/ no Peak-to-peak | Optimized EPAP w/ Max Peak-to-peak | Non-optimized EPAP w/ no Peak-to-peak
Number analyzed (Participants) | 2 | 2 | 2 | 2
mL/min | 6708 (492) | 5906.5 (168.5) | 6791 (1184) | 6072 (576)

ADVERSE EVENTS:
Time Frame: 10 days
Groups:
- Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized P2P: Optimal - optimal EPAP determination first, Optimized P2P - Optimized EPAP w/ max peak-to-peak second, Non-Optimized NP2P - Non-Optimized EPAP w/ no peak-to-pea third, and Optimized P2P - optimized EPAP w/ peak-to-peak last
Arm/Group | Screening Period | Optimal, Optimized P2P, Non-Optimized NP2P, Optimized NP2P | Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized P2P
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Period (N=10) | Optimal, Optimized P2P, Non-Optimized NP2P, Optimized NP2P (N=2) | Optimal, Optimized NP2P, Non-Optimized NP2P, Optimized P2P (N=1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to low enrollment.

Washout period between sessions of 20-30 minutes was not sufficient for CO2 to return to baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No